CLINICAL TRIAL: NCT06656858
Title: The Acute Effects of Static and PNF Stretching Exercise With Blood Flow Restriction on Hamstring Flexibility, Muscle Strength and Single Leg Hop in Athletes : A Randomized Controlled Trial
Brief Title: The Acute Effects of Static and PNF Stretching Exercise With Blood Flow Restriction in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ayşe Birsu Topcugil Kırık, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5016-GOA
Record Dates: First submitted 2024-02-19; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Athletes
Keywords: blood flow restriction, stretching, flexibility, hamstring
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Static stretching (Active Comparator): Static stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds.
  Interventions: Other: Static stretching
- PNF stretching (Active Comparator): PNF stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds.
  Interventions: Other: PNF stretching
- Static stretching with BFR (Experimental): Static stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds with BFR application.
  Interventions: Other: Static stretching with BFR
- PNF stretching with BFR (Experimental): PNF stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds with BFR application
  Interventions: Other: PNF stretching with BFR
- Control (Other): No stretching was applied to the control group. An information brochure about hamstring injuries was provided to the participants.
  Interventions: Other: Control

INTERVENTIONS:
Other: Static stretching — Static stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds
  Arms: Static stretching
Other: PNF stretching — PNF stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds.
  Arms: PNF stretching
Other: Static stretching with BFR — Static stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds with BFR application.
  Arms: Static stretching with BFR
Other: PNF stretching with BFR — PNF stretching exercises were performed on the dominant leg's hamstring muscle group for 3 sets of 15 seconds with BFR application.
  Arms: PNF stretching with BFR
Other: Control — No stretching was applied to the control group. An information brochure about hamstring injuries was provided to the participants.
  Arms: Control

SUMMARY:
The study aims to examine the acute effects of static and proprioceptive neuromuscular facilitation stretching exercises with blood flow restriction on hamstring flexibility, muscle strength, and single leg hop in athletes. Outcome measures were hip range of motion, isometric and eccentric hamstring muscle strength, and single leg hop distance.

DETAILED DESCRIPTION:
A total of 109 athletes were included in the study. Participants were randomized into five groups: (1) static stretching, (2) proprioceptive neuromuscular facilitation (PNF) stretching, (3) blood flow restriction (BFR) + static stretching, (4) BFR + PNF stretching, and (5) control groups. Stretching exercises were performed on the dominant leg hamstring muscle group for 3 sets of 15 seconds each. BFR was applied during the stretching to the blood flow restriction (BFR) + static stretching and BFR + PNF stretching groups. No stretching was applied to the control group.

Assessments were performed at baseline and immediately after stretching. Hamstring flexibility (hip joint range of motion) was assessed via the passive straight leg raise test. Isometric and eccentric hamstring muscle strength were measured using a hand-held dynamometer, and muscle power was assessed using the single leg hop distance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years old
* Engaged in regular physical activity for at least 8 hours a week for the last 6 months
* Body mass index (BMI) < than 30 kg/m²
* Momentary blood pressure less than 135/85 mmHg

Exclusion Criteria:

* History of fractures or surgical operations involving the lower limbs, hips, or lumbar region
* history of fractures, surgeries and other diagnosed medical conditions on the lower extremity, hip, and lumbar region
* Systemic musculoskeletal disease
* Pain in the lower back, hips, or lower extremities
* Known hip deformity or diagnosis of scoliosis
* History of deep vein thrombosis or embolism
* Diagnosis of circulatory system diseases such as hypertension or peripheral vascular disease
* History of anemia
* Previous cerebrovascular disease or myocardial infarction.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
hamstring flexibility | immediately after intervention
  Passive straight leg rise test for dominant leg

SECONDARY OUTCOMES:
Power | immediately after intervention
  single leg hop distance for dominant and non-dominant leg
muscle strength | immediately after intervention
  isometric and eccentric hamstring muscle strength of the dominant leg

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Birsu Topcugil Kirik, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Sports Medicine Department, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No